CLINICAL TRIAL: NCT05487625
Title: Effects of Narratives on Demand for Low and High Ventilated Cigarettes and Substitution for Alternative Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: University of Minnesota (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roberta Freitas-Lemos, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB #22-432; 5P01CA217806 (NIH)
Record Dates: First submitted 2022-07-31; First posted 2022-08-04 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Commerce

STUDY DESIGN:
Intervention Model Description: Participants will complete five ETM conditions, which include six trials assessing different cigarette prices: a) high-ventilated cigarette alone, b) low-ventilated cigarette alone, c) high- and low-ventilated cigarette with high-ventilated cigarettes increasing in price, d) high- and low-ventilated cigarette with low-ventilated cigarettes increasing in price, and e) usual, high- and low-ventilated cigarette with usual cigarettes increasing in price.
Who Masked: Participant
Masking Description: Participants will be provided with study cigarettes (commercially available) however the brand will not be provided to them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Narratives (Experimental): High-ventilated cigarette smokers will be exposed to a narrative about the negative consequences of smoking ventilated cigarettes and all of the conditions described in the intervention section.
  Interventions: Behavioral: High-ventilated cigarette alone; Behavioral: Low-ventilated cigarette alone; Behavioral: High- and low-ventilated cigarette with high-ventilated cigarettes increasing in price; Behavioral: Low- and high-ventilated cigarette with high-ventilated cigarettes increasing in price; Behavioral: Usual, high- and low-ventilated cigarette with usual cigarettes increasing in price.
- Fact sheet (Experimental): High-ventilated cigarette smokers will be exposed to fact sheet about the negative consequences of smoking ventilated cigarettes and all of the conditions described in the intervention section.
  Interventions: Behavioral: High-ventilated cigarette alone; Behavioral: Low-ventilated cigarette alone; Behavioral: High- and low-ventilated cigarette with high-ventilated cigarettes increasing in price; Behavioral: Low- and high-ventilated cigarette with high-ventilated cigarettes increasing in price; Behavioral: Usual, high- and low-ventilated cigarette with usual cigarettes increasing in price.
- Control (Experimental): High-ventilated cigarette smokers will be not be exposed to any messages and will complete all of the conditions described in the intervention section.
  Interventions: Behavioral: High-ventilated cigarette alone; Behavioral: Low-ventilated cigarette alone; Behavioral: High- and low-ventilated cigarette with high-ventilated cigarettes increasing in price; Behavioral: Low- and high-ventilated cigarette with high-ventilated cigarettes increasing in price; Behavioral: Usual, high- and low-ventilated cigarette with usual cigarettes increasing in price.

INTERVENTIONS:
Behavioral: High-ventilated cigarette alone — High-ventilated cigarettes are the only available cigarettes in the Experimental Tobacco Marketplace which increases in price across trials. Other nicotine/tobacco products are available in the Experimental Tobacco Marketplace at market price. Note that all participants will complete all the specified conditions.
Behavioral: Low-ventilated cigarette alone — Low-ventilated cigarettes are the only available cigarettes in the Experimental Tobacco Marketplace which increases in price across trials. Other nicotine/tobacco products are available in the Experimental Tobacco Marketplace at market price. Note that all participants will complete all the specified conditions.
Behavioral: High- and low-ventilated cigarette with high-ventilated cigarettes increasing in price — High- and low ventilated cigarettes are available in the Experimental Tobacco Marketplace with high-ventilated cigarettes increasing in price across trials. Other nicotine/tobacco products are available in the Experimental Tobacco Marketplace at market price. Note that all participants will complete all the specified conditions.
Behavioral: Low- and high-ventilated cigarette with high-ventilated cigarettes increasing in price — Low- and high-ventilated cigarettes are available in the Experimental Tobacco Marketplace with low-ventilated cigarettes increasing in price across trials. Other nicotine/tobacco products are available in the Experimental Tobacco Marketplace at market price. Note that all participants will complete all the specified conditions.
Behavioral: Usual, high- and low-ventilated cigarette with usual cigarettes increasing in price. — Usual cigarette, low- and high-ventilated cigarettes are available in the Experimental Tobacco Marketplace with usual cigarettes increasing in price across trials. Other nicotine/tobacco products are available in the Experimental Tobacco Marketplace at market price. Note that all participants will complete all the specified conditions.

SUMMARY:
This study will investigate the effects of narratives on demand for low and high ventilated cigarettes and substitution for alternative products in the Experimental Tobacco Marketplace.

DETAILED DESCRIPTION:
An important aim of tobacco control is to reduce demand for the most harmful products. One product feature that could be changed to benefit public health is cigarette filter ventilation. A recent review examined the effects of cigarette filter ventilation and concluded that filter ventilation, by changing how a cigarette burns, yields more mutagens and carcinogens, and results in greater puff volume and possibly depth of inhalation, which has led to increases in peripheral lung adenocarcinomas. This study will use a novel method, the Experimental Tobacco Marketplace (ETM), to compare the impact of a narrative and a factsheet on the negative consequences of filter ventilation on tobacco product purchases. High-ventilated cigarette smokers will complete multiple scenarios in the ETM.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Be at least 21 years of age or older
* Provide a breath sample for measuring carbon monoxide (CO ≥ 8 ppm)
* Stable tobacco use patterns for at least three months
* Be willing to sample the study cigarettes (high- and low-ventilated cigarettes)
* Report smoking a high-ventilated cigarette (>= 20% ventilation)
* Report smoking at least 10 cigarettes per day

Exclusion Criteria:

* Have plans to move out of the area
* Have a serious or unstable physical or mental health condition
* Taking a tobacco cessation medication or medication that interferes with nicotine metabolism, motivation or reinforcement
* Report concrete, immediate plans to alter/quit using their usual nicotine products at the beginning of the study

Note: Participants may be withdrawn from the study after providing consent if they submit an invalid breath sample (CO ≥ 8 ppm).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren K Bickel, Ph.D., Principal Investigator — Fralin Biomedical Research Institute at VTC
Locations (1):
- Addiction recovery Research center, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
The study team will share de-identified data upon request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Narratives: High-ventilated cigarette (HVC) smokers will be exposed to a narrative about the negative consequences of smoking HVC and all of the conditions described in the intervention section.
  HVC alone: HVC are the only available cigarettes in the ETM which increases in price across trials. Other products are available in the ETM at market price (MP). Note that all participants will complete all the specified conditions.
  Low-ventilated cigarette (LVC) alone: LVC are the only available cigarettes in the ETM which increases in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
  HVC and LVC with HVC increasing in price: HVC and LVC are available in the ETM with HVC increasing in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
  LVC and HVC with HVC increasing in price: LVC and HVC are available in the ETM with LVC increasing in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
  Usual, HVC and LVC with usual cigarettes increasing in price.: Usual cigarette, HVC and LVC are available in the ETM with usual cigarettes increasing in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
- Fact Sheet: High-ventilated cigarette (HVC) smokers will be exposed to fact sheet about the negative consequences of smoking ventilated cigarettes and all of the conditions described in the intervention section.
  HVC alone: HVC are the only available cigarettes in the ETM which increases in price across trials. Other products are available in the ETM at market price (MP). Note that all participants will complete all the specified conditions.
  Low-ventilated cigarette (LVC) alone: LVC are the only available cigarettes in the ETM which increases in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
  HVC and LVC with HVC increasing in price: HVC and LVC are available in the ETM with HVC increasing in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
  LVC and HVC with HVC increasing in price: LVC and HVC are available in the ETM with LVC increasing in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
  Usual, HVC and LVC with usual cigarettes increasing in price.: Usual cigarette, HVC and LVC are available in the ETM with usual cigarettes increasing in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
- Control: High-ventilated cigarette (HVC) smokers will be not be exposed to any messages and will complete all of the conditions described in the intervention section.
  HVC alone: HVC are the only available cigarettes in the ETM which increases in price across trials. Other products are available in the ETM at market price (MP). Note that all participants will complete all the specified conditions.
  Low-ventilated cigarette (LVC) alone: LVC are the only available cigarettes in the ETM which increases in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
  HVC and LVC with HVC increasing in price: HVC and LVC are available in the ETM with HVC increasing in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
  LVC and HVC with HVC increasing in price: LVC and HVC are available in the ETM with LVC increasing in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
  Usual, HVC and LVC with usual cigarettes increasing in price.: Usual cigarette, HVC and LVC are available in the ETM with usual cigarettes increasing in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
Period: Overall Study
Arm/Group | Narratives | Fact Sheet | Control
Started | 28 | 30 | 29
HVC Alone | 27 | 28 | 27
LVC Alone | 27 | 28 | 27
HVC and LVC With HVC Increasing in Price | 27 | 28 | 27
LVC and HVC With HVC Increasing in Price | 27 | 28 | 27
Usual, HVC and LVC With Usual Cigarettes Increasing in Price | 27 | 28 | 27
Completed | 27 | 28 | 27
Not Completed | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Narratives | Fact Sheet | Control | Total
Number analyzed (Participants) | 27 | 28 | 27 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years of age] | 46.37 (10.76) | 40.32 (10.06) | 43.81 (7.71) | 43.46 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 19 | 50
  Male | 11 | 13 | 8 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 28 | 27 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 1 | 4
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 2 | 7 | 15
  White | 20 | 22 | 19 | 61
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Fagerstrom Test for Cigarette Dependence [Mean (Standard Deviation); unit: Scores on a scale] — The Fagerstrom Test for Cigarette Dependence is a 6-item scale to assess cigarette dependence. Scores range from 0 to 10: 0 represents no dependence, 1-2 low dependence, 3-4 low to moderate dependence, 5-7 moderate dependence and 8-10 represents high dependence. We summed all participants scores and calculated the mean for each group as well as the standard deviation.
  Scores on a scale | 5.52 (2.19) | 6.25 (2.03) | 5.26 (1.58) | 5.68 (1.97)

OUTCOME MEASURES:

1. Primary Outcome: Nicotine/Tobacco Products Substitution Intercept
Description: Participants completed purchasing trials in an Experimental Tobacco Marketplace (ETM), where cigarette prices increased (type varied by condition) while other product prices remained at market value. The extent to which other nicotine/tobacco products substituted for usual, high-, and low-ventilated cigarettes was assessed. The quantity of products purchased in the ETM was converted to milligrams (mg) of nicotine to standardize the unit of measurement across products. The data reflect the relationship between nicotine purchased (mg; y-axis) and cigarette price (x-axis).
  To obtain estimates of substitution of price-constant products in the different ETM conditions, the investigators used ordinary least squares regression to predict total mg of nicotine purchased of the price constant product. Y-intercept of price-constant products is reported.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: Mg of Nicotine purchased
Groups:
- Narratives: High-ventilated cigarette (HVC) smokers will be exposed to a narrative about the negative consequences of smoking ventilated cigarettes and all of the conditions described in the intervention section.
  HVC alone: HVC are the only available cigarettes in the ETM which increases in price across trials. Other products are available in the ETM at market price (MP). Note that all participants will complete all the specified conditions.
  Low-ventilated cigarette (LVC) alone: LVC are the only available cigarettes in the ETM which increases in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
  HVC and LVC with HVC increasing in price: HVC and LVC are available in the ETM with HVC increasing in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
  LVC and HVC with HVC increasing in price: LVC and HVC are available in the ETM with LVC increasing in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
  Usual, HVC and LVC with usual cigarettes increasing in price.: Usual cigarette, HVC and LVC are available in the ETM with usual cigarettes increasing in price across trials. Other products are available in the ETM at MP. Note that all participants will complete all the specified conditions.
Arm/Group | Narratives | Fact Sheet | Control
Number analyzed (Participants) | 27 | 28 | 27
Mg of Nicotine purchased
  High-ventilated cigarette alone: e-cigarette estimated intercept | 16.4 (37.6) | 94.2 (36.9) | 47.8 (37.5)
  Low-ventilated cigarette alone: e-cigarette estimated intercept | 56.0 (43.5) | 12.1 (42.8) | 67.4 (43.5)
  HVC and LVC cigarette with HVC cigarettes increasing in price: LVC estimated intercept | 129.8 (48.6) | 182.0 (47.9) | 236.2 (48.6)
  HVC and LVC cigarette with HVC cigarettes increasing in price: e-cigarette estimated intercept | 49.9 (48.6) | 56.9 (47.9) | 30.2 (48.6)
  HVC and LVC cigarette with LVC cigarettes increasing in price: e-cigarette estimated intercept | 56.1 (45.4) | 40.3 (44.8) | 40.7 (45.4)
  HVC and LVC cigarette with LVC cigarettes increasing in price: HVC estimated intercept | 102.3 (45.4) | 184.8 (44.8) | 206.9 (45.4)
  Usual, HVC and LVC cigarette with usual cigarettes increasing in price: e-cigarette intercept | 59.43 (37.9) | 40.35 (37.4) | 2.80 (37.9)
  Usual, HVC and LVC cigarette with usual cigarettes increasing in price: HVC intercept | -55.80 (37.9) | -24.32 (37.4) | 35.66 (37.9)
  Usual, HVC and LVC cigarette with usual cigarettes increasing in price: LVC intercept | 6.24 (37.9) | 23.99 (37.4) | -5.20 (37.9)

2. Primary Outcome: Cigarette Demand Intensity q0
Description: Participants completed purchasing trials in an Experimental Tobacco Marketplace (ETM), where cigarette prices increased (type varied by condition) while other product prices remained at market value. The extent to which other nicotine/tobacco products substituted for usual, high-, and low-ventilated cigarettes was assessed. The quantity of products purchased in the ETM was converted to milligrams (mg) of nicotine to standardize the unit of measurement across products. The data reflect the relationship between nicotine purchased (mg; y-axis) and cigarette price (x-axis). Demand was estimated using the exponential equation: Q = Q0 * 10^k(exp(-αQ0C) - 1), where Q is nicotine purchased (mg), C is price, Q0 is demand intensity (purchases at no cost), k is the function's logarithmic span, and α is demand elasticity. Intensity q0 is reported, which represents the estimated mg of nicotine purchased when cigarettes are free (price = 0).
Time Frame: 1 day
Measure: Mean (Standard Error); unit: Mg of Nicotine purchased
Arm/Group | Narratives | Fact Sheet | Control
Number analyzed (Participants) | 27 | 28 | 27
Mg of Nicotine purchased
  Cigarette demand intensity q0: usual | 2509.951 (636.7094) | 2446.043 (629.3318) | 2002.901 (431.5768)
  Cigarette demand intensity q0: HVC and LVC with HVC increasing in price | 1226.371 (313.1189) | 1389.097 (376.9664) | 1201.065 (333.2428)
  Cigarette demand intensity q0: LVC and HVC with LVC increasing in price | 1296.955 (371.9530) | 1106.049 (292.4133) | 1393.520 (416.9316)
  Cigarette demand intensity q0: HVC only | 1293.099 (247.6387) | 2207.993 (483.5283) | 1395.041 (321.9870)
  Cigarette demand intensity q0: LVC only | 2289.174 (613.9061) | 1379.648 (215.8875) | 2085.754 (565.8513)

3. Primary Outcome: Nicotine/Tobacco Products Substitution Slope
Description: Participants completed purchasing trials in an Experimental Tobacco Marketplace (ETM), where cigarette prices increased (type varied by condition) while other product prices remained at market value. The extent to which other nicotine/tobacco products substituted for usual, high-, and low-ventilated cigarettes was assessed. The quantity of products purchased in the ETM was converted to milligrams (mg) of nicotine to standardize the unit of measurement across products. The data reflect the relationship between nicotine purchased (mg; y-axis) and cigarette price (x-axis).
  To obtain estimates of substitution of price-constant products in the different ETM conditions, the investigators used ordinary least squares regression to predict total mg of nicotine purchased of the price-constant product. Slope of price-constant products is reported, which represents the change in mg of nicotine purchased of price-constant products divided by the change in cigarette price.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: Mg of nicotine/price US$
Arm/Group | Narratives | Fact Sheet | Control
Number analyzed (Participants) | 27 | 28 | 27
Mg of nicotine/price US$
  High-ventilated cigarette alone: e-cigarette estimated slope | 13.24 (8.35) | -10.33 (8.24) | 1.96 (8.35)
  Low-ventilated cigarette alone: e-cigarette tobacco estimated slope | 1.65 (9.47) | 11.50 (9.34) | -4.26 (9.47)
  HVC and LVC cigarette with HVC cigarettes increasing in price: LVC estimated slope | 26.48 (9.89) | 20.94 (9.79) | 27.70 (9.89)
  HVC and LVC cigarette with HVC cigarettes increasing in price: e-cigarette estimated slope | 1.88 (9.89) | -3.67 (9.79) | 3.09 (9.89)
  HVC and LVC cigarette with LVC cigarettes increasing in price: e-cigarette estimated slope | 0.989 (9.65) | 1.593 (9.54) | 0.110 (9.65)
  HVC and LVC cigarette with LVC cigarettes increasing in price: HVC estimated slope | 24.678 (9.65) | 25.283 (9.54) | 23.800 (9.65)
  Usual, HVC and LVC cigarette with usual cigarettes increasing in price: e-cigarette slope | -4.370 (8.17) | -0.643 (8.09) | 7.577 (8.17)
  Usual, HVC and LVC cigarette with usual cigarettes increasing in price: HVC slope | 28.306 (8.17) | 32.033 (8.09) | 40.253 (8.17)
  Usual, HVC and LVC cigarette with usual cigarettes increasing in price: LVC slope | 20.456 (8.17) | 24.182 (8.09) | 32.403 (8.17)

4. Primary Outcome: Cigarette Demand Elasticity Alpha
Description: Participants completed purchasing trials in an Experimental Tobacco Marketplace (ETM), where cigarette prices increased (type varied by condition) while other product prices remained at market value. The extent to which other nicotine/tobacco products substituted for usual, high-, and low-ventilated cigarettes was assessed. The quantity of products purchased in the ETM was converted to milligrams (mg) of nicotine to standardize the unit of measurement across products. The data reflect the relationship between nicotine purchased (mg; y-axis) and cigarette price (x-axis). Demand was estimated using the exponential equation: Q = Q0 * 10^k(exp(-αQ0C) - 1), where Q is nicotine purchased (mg), C is price, Q0 is demand intensity (purchases at no cost), k is the function's logarithmic span, and α is demand elasticity. Elasticity alpha is reported, which represents the sensitivity of purchasing to changes in cigarette price.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: Mg of Nicotine purchased/Price changes
Arm/Group | Narratives | Fact Sheet | Control
Number analyzed (Participants) | 27 | 28 | 27
Mg of Nicotine purchased/Price changes
  Cigarette demand elasticity alpha: usual | 0.0001184530 (0.00002668313) | 0.0001866522 (0.00005510821) | 0.0006728454 (0.0004281379)
  Cigarette demand elasticity alpha: HVC and LVC with HVC increasing in price | -0.004862780 (0.00730483) | 0.003933976 (0.00373252) | 0.002001107 (0.00192290)
  Cigarette demand elasticity alpha: LVC and HVC with LVC increasing in price | 0.0001730126 (0.00008899978) | 0.0010937345 (0.0007710276) | 0.0004953039 (0.0003009148)
  Cigarette demand elasticity alpha: HVC only | 0.005474398 (0.002837352) | 0.002718229 (0.002489950) | 0.006274115 (0.005146063)
  Cigarette demand elasticity alpha: LVC only | 0.0017715209 (0.0015139344) | 0.0003113996 (0.0001296562) | 0.0058833919 (0.0053767638)

ADVERSE EVENTS:
Time Frame: Approximately 2-3 weeks.
Description: Adverse events were assessed in a systematic manner. Specifically, this adverse event was identified before the intervention phase, during the period when a participant was sampling products at home. The participant reported experiencing withdrawal symptoms after using the products.
Arm/Group | Narratives | Fact Sheet | Control
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 1/28 | 0/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Narratives (N=27) | Fact Sheet (N=28) | Control (N=27)
Gastrointestinal Issues (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — You might experience adverse effects associated with the use of nicotine products (e.g., nausea, vomiting, dizziness, diarrhea, weakness, and rapid heartbeat).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT05487625/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT05487625/SAP_001.pdf
  • Informed Consent Form (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT05487625/ICF_002.pdf